CLINICAL TRIAL: NCT05985200
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Rising Intravenous Doses of BI 3032950 in Healthy Male and Female Subjects (Single-blind, Randomised Within Dose Groups, Placebo-controlled Parallel-group Design)
Brief Title: A Study in Healthy People to Test How Well Repeated Doses of BI 3032950 Are Tolerated
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1486-0002; U1111-1289-1904 (Registry Identifier: WHO Registry); 2023-503332-40-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- BI 3032950: Dose group 1 (Experimental)
  Interventions: Drug: BI 3032950
- BI 3032950: Dose group 2 (Experimental)
  Interventions: Drug: BI 3032950
- BI 3032950: Dose group 3 (Experimental)
  Interventions: Drug: BI 3032950
- BI 3032950: Dose group 4 (Experimental)
  Interventions: Drug: BI 3032950
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo matching BI 3032950

INTERVENTIONS:
Drug: BI 3032950 — BI 3032950
  Arms: BI 3032950: Dose group 1; BI 3032950: Dose group 2; BI 3032950: Dose group 3; BI 3032950: Dose group 4
Drug: Placebo matching BI 3032950 — Placebo matching BI 3032950
  Arms: Placebo

SUMMARY:
The main objectives of this trial are to investigate safety, tolerability, pharmacokinetics and pharmacodynamics following multiple rising intravenous doses of BI 3032950 in healthy male subjects and postmenopausal or surgically sterilised female subjects (women not of child bearing potential (WNOCBP)).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects and female subjects not of child bearing potential (women not of child bearing potential (WNOCBP)) - postmenopausal or surgically sterilised female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
2. Age of 18 to 65 years (inclusive)
3. Body mass index (BMI) of 18.5 to 29.9 kg/m^2 (inclusive)
4. Signed and dated written informed consent in accordance with International conference on harmonisation-good clinical practice (ICH-GCP) and local legislation prior to admission to the trial
5. Male subjects (including male subjects with pregnant partners) who meet any of the criteria listed in the protocol for a highly effective contraception from the first administration of trial medication until the end of study (EoS) visit.
6. Postmenopausal or surgically sterilised female subjects (WNOCBP) who are:

   * Confirmed surgically sterilised (including hysterectomy, bilateral salpingectomy and bilateral oophorectomy), or
   * Postmenopausal, defined as at least 1 year of spontaneous amenorrhea without an alternative medical cause Further inclusion criteria apply.

Exclusion Criteria:

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 100 beats per minute (bpm); in case of documented 'white coat hypertension' the decision for eligibility is left to the investigator
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator Further exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
Occurrence of any treatment-emergent adverse event | Up to Day 137

SECONDARY OUTCOMES:
Occurrence of any treatment-emergent adverse event assessed as drug-related by the investigator | Up to Day 137
Area under the concentration-time curve of the analyte in serum over a uniform dosing interval τ (AUCτ,) | From Day 22 to Day 134
Maximum measured concentration of the analyte in serum (Cmax) | From Day 22 to Day 134

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Life Science Services - Clinical Research, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency.

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com